CLINICAL TRIAL: NCT02262429
Title: Does a Rapid, Comprehensive Oral Nutritional Supplementation Quality Improvement Program (QIP) Reduce 30-Day Readmission in Malnourished Hospitalized Patients?
Brief Title: Quality Improvement Program (QIP) to Reduce 30-Day Readmission in Malnourished Hospitalized Patients
Status: Terminated | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: HA13
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ONS QIP: Two (2) hospitals will administer the new rapid, comprehensive oral nutritional supplementation (ONS) QIP.
  Interventions: Other: ONS QIP
- ONS Standard Feeding: Two (2) hospitals will use their current "standard" ONS feeding protocol.
  Interventions: Other: ONS Standard Feeding

INTERVENTIONS:
Other: ONS QIP — Rapid comprehensive ONS, dietary consult, follow up phone calls
  Groups: ONS QIP
Other: ONS Standard Feeding — Standard of care
  Groups: ONS Standard Feeding

SUMMARY:
Newly admitted patients will be screened for risk of malnutrition. Patients will receive either the feeding protocol or current oral nutrition supplement (ONS) practice, pending location. Patients will continue the nutrition plan taking the supplement post discharge. Study team will follow-up with telephone calls to help support post-discharge ONS compliance. Quality and service utilization data will be gathered for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age.
* Patient is screened for malnutrition with an MST score ≥ 2 (see Appendix C).
* Patient has length of stay of hospital stay > 2 days.
* Patient is able to consume foods and beverages orally.
* Patient receives Ensure, Nepro or Glucerna during the course of his or her hospital stay in connection with the QIP.

Exclusion Criteria:

* Patient is pregnant.
* Patient is intubated, receiving tube feeding or parenteral nutrition.
* Patient unable to provide HIPAA authorization and informed consent.
* Patient is discharged to hospice care.
* Patient has a condition that would preclude ingestion / absorption of the oral nutritional supplements, including allergic response to any ONS ingredient.
* Patient has severe dementia or delirium, brain metastases, eating disorder, history of significant neurological or psychiatric disorder.
* Patient has stated an allergy or intolerance to any of the ingredients in the study products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly admitted patients to four hospitals within the Advocate Health Care System that have been identifed to be at risk for malnutrition.
Sampling Method: Non-Probability Sample
Enrollment: 2386 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Post-discharge readmissions | November 2014 - April 2015, 30 days post discharge
  Non-elective readmission 30 days post discharge.

SECONDARY OUTCOMES:
Hospital length of stay | October 2014 - March 2015, up to 6 months
  Length of stay in the hospital will be calculated by looking at the admission and discharge dates.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Partridge, PhD, MBA, Study Director — Abbott Nutrition
Locations (4):
- United States (4):
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois

REFERENCES:
- [Derived] Sriram K, Sulo S, VanDerBosch G, Kozmic S, Sokolowski M, Summerfelt WT, Partridge J, Hegazi R, Nikolich S. Nutrition-Focused Quality Improvement Program Results in Significant Readmission and Length of Stay Reductions for Malnourished Surgical Patients. JPEN J Parenter Enteral Nutr. 2018 Aug;42(6):1093-1098. doi: 10.1002/jpen.1040. Epub 2018 Feb 2. PMID 29392736